CLINICAL TRIAL: NCT07310368
Title: Comparison of the Effectiveness of Mobilization and Myofascial Release Techniques on Pain, Postural Control, and Spinal Mobility in Patients With Sacroiliac Joint Dysfunction
Brief Title: Comparison of the Effectiveness of Mobilization and Myofascial Release Techniques in Patients With Sacroiliac Joint Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Safak Kuzu, Assist. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52066301980*
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroiliac Joint Dysfunction; Mobilization; myofascial release

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release (Experimental): The myofascial release time for each muscle was 90 to 120 seconds, applied twice per session. 1. Myofascial release of the erector spinae muscles: the patient assumed a prone position; and the therapist stood at the patient's pelvis on the treatment side, applying the cross-hand technique. 2. Myofascial release of the quadratus lumborum muscle and thoracolumbar fascia: to increase the stretching force on the muscle, the patient lay on their side on the untreated side and placed a pillow under their lower back. The therapist stood behind the patient at the level of the patient's pelvis, applying the cross-hand technique. 3. Myofascial release of the piriformis muscle: The patient assumed a lateral recumbent position with the treated side on top. To increase muscle tension, the upper lower extremity was placed in hip flexion and adduction in front of the patient's lower extremity.
  Interventions: Other: Traditional treatment program; Other: myofascial relaxation
- Mobilization (Experimental): Patients lay on their side with the sacroiliac joint restricted at the top, and sacroiliac manipulation was performed. Then, the physiotherapist flexed the lumbar spine by moving toward the upper part of the thigh, applying an impulse using the intermittent stretching technique in the direction of the major thoracanthus from the iliac crest. In the prone position, caudal traction, traction of the sacrum relative to the ilium, and traction stretches from the iliac crests will be applied.
  Interventions: Other: Traditional treatment program; Other: Mobilization

INTERVENTIONS:
Other: Traditional treatment program — Bridge exercises, back extension exercises, and sit-up exercises as strengthening exercises. These exercises will be preferred to strengthen the abdominal and back muscles. Ultrasound will be applied to the sacroiliac region in the prone position. The practitioner will rotate the ultrasound head in a circular motion at a 90-degree angle to apply ultrasound to the right and left sacroiliac joints. A 4 cm wide probe will be used to apply continuous ultrasound at 1 MHz and 1.5 watts/cm2 for 8 minutes.
Other: myofascial relaxation — The myofascial release time for each muscle was 90 to 120 seconds, applied twice per session. 1. Myofascial release of the erector spinae muscles: the patient assumed a prone position; and the therapist stood at the patient's pelvis level on the treatment side, applying the cross-hand technique. 2. To increase muscle tension, the patient's lower extremity was placed in hip flexion and adduction at the highest point. The therapist stood behind the patient, at the level of the patient's pelvis, and applied the transverse tapping technique using the knuckles. 4. Myofascial release of the gluteus medius muscle: The patient assumed a lateral recumbent position on the untreated side. The therapist stood behind the patient, at the level of the patient's pelvis, and applied the vertical tapping technique using the knuckles.
  Arms: Myofascial Release
Other: Mobilization — Patients lay on their side with the sacroiliac joint restricted at the top, and sacroiliac manipulation was performed. Then, the physiotherapist flexed the lumbar spine by moving toward the upper part of the thigh, applying an impulse using the intermittent stretching technique in the direction of the major thoracanthus from the iliac crest. In the prone position, caudal traction, traction of the sacrum relative to the ilium, and traction stretches from the iliac crests will be applied.
  Arms: Mobilization

SUMMARY:
Sacroiliac joint dysfunction (SIED) is one of the major causes of chronic mechanical low back pain and is associated with pain, postural control impairment, and functional limitations. While manual therapy approaches are commonly used in the treatment of sacroiliac joint pain, evidence regarding the clinical superiority of different manual techniques is limited.

This study was designed as a prospective, randomized controlled trial to compare the effects of myofascial release techniques and sacroiliac joint mobilizations, applied in addition to a traditional physical therapy program, on pain intensity, spinal mobility, postural control, and functional status in women diagnosed with sacroiliac joint dysfunction.

The study plans to include female individuals aged 18-65 years with a Visual Analog Scale (VAS) score ≥3 who have been diagnosed with sacroiliac joint dysfunction according to international diagnostic criteria. Participants will be randomly assigned to two groups: one group will receive traditional treatment combined with myofascial release techniques, while the other group will receive traditional treatment combined with sacroiliac joint mobilizations. Interventions will be performed three days per week for six weeks.

Primary and secondary outcome measures will include pain intensity (VAS), postural control (Biodex Balance System), spinal mobility, and postural endurance (Spinal Mouse) assessments. Participants will be randomly assigned to two groups: one group will receive traditional treatment combined with myofascial release techniques, while the other group will receive traditional treatment combined with sacroiliac joint mobilizations. Interventions will be performed three days a week for six weeks.

Primary and secondary outcome measures will include pain intensity (VAS), postural control (Biodex Balance System), spinal mobility, and postural endurance (Spinal Mouse) assessments. All assessments will be conducted before treatment and at the end of the six-week intervention period.

This study aims to provide clinical evidence regarding the comparative effectiveness of manual therapy approaches in the conservative treatment of sacroiliac joint dysfunction and to contribute to clinical decision-making processes.

DETAILED DESCRIPTION:
This study is a clinical prospective, randomized controlled trial evaluating two different manual therapy approaches added to a traditional physical therapy program in women diagnosed with sacroiliac joint dysfunction (SIED). The primary objective of the study is to comparatively evaluate the effects of myofascial release techniques and sacroiliac joint mobilizations on pain, spinal mobility, postural control, and postural endurance.

Eligible participants included in the study will be randomly assigned to two intervention groups using a computer-based randomization method. Both groups will receive the same traditional physical therapy program three days a week for six weeks. This approach aims to ensure that any differences between the groups are solely attributable to the manual therapy technique applied.

The traditional physical therapy program will include stabilization and strengthening exercises targeting the abdominal and back muscles (bridge, back extension, and sit-up exercises) and therapeutic ultrasound application to the sacroiliac region. This program will be applied to all participants for the same duration and intensity.

Myofascial release techniques will be used in addition to the traditional physical therapy program. The myofascial release techniques applied in this group will be planned to target the erector spinae, quadratus lumborum, thoracolumbar fascia, piriformis, and gluteus medius muscles. The applications will be performed in accordance with the principles of soft tissue mobilization and fascial release.

Mobilization will be treated with sacroiliac joint mobilization techniques in addition to the traditional physical therapy program. In this group, posterior-anterior and inferior mobilization techniques will be applied to regulate the biomechanics of the sacroiliac joint and increase joint mobility. Mobilizations will be graded according to the patient's tolerance and performed within safe limits.

All interventions will be performed by physical therapists experienced in manual therapy. Participants will not be allowed to receive any other manual therapy or alternative treatment during the treatment period.

Outcome assessments will be conducted before the treatment program (baseline) and at the end of the six-week intervention period. Pain intensity will be assessed using the Visual Analog Scale (VAS) as the primary outcome measure. Secondary outcome measures will include postural control (Biodex Balance System), spinal mobility, and postural endurance (Spinal Mouse system). All measurements will be performed by the same evaluator under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Being a female individual between the ages of 18 and 65.
* Having been diagnosed with sacroiliac joint dysfunction (according to the International Association for the Study of Pain criteria).
* Having localized pain in the sacroiliac joint region and pain that may radiate to the hip, groin, or lower extremities.
* Positivity in at least 3 out of 5 sacroiliac joint-specific provocation tests (Vorlauf, Gillet, irritation point positivity, posterior shear test, compression test).
* Pain intensity of ≥3 as assessed by the Visual Analog Scale (VAS).
* Volunteering to participate in the study and providing written informed consent.

Exclusion Criteria:

* History of surgery involving the spine, pelvis, or lower extremities.
* Presence of lumbar disc herniation, spinal stenosis, or acute pathologies of the hip joint.
* Diagnosis of piriformis syndrome or low back/hip pain originating from sources other than the sacroiliac joint.
* Known central or peripheral nervous system disease or progressive neurological deficit.
* History of rheumatological disease (rheumatoid arthritis, ankylosing spondylitis, etc.).
* Pregnancy or the presence of a serious systemic disease that could prevent participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Postural control assessment | 6 week
  Postural control will be assessed statically and dynamically. The Biodex balance system (Biodex Medical System Inc., NY, USA, SW45 30D E6N Model, SD 950 304) will be used. This device creates stability indices by evaluating movements in the overall, anterior-posterior, and medial-lateral directions. For static balance assessment, the subject is asked to hold a small circle containing a black dot representing their center of gravity without moving it for 20 seconds, repeated 3 times. For dynamic assessment, the floor movement level is set to 12 at the start and gradually reduced to 9 throughout the test. At these levels, the subject attempts to keep their center of gravity balanced within the small circle. Total, anterior-posterior (A-P), and medial-lateral (M-L) values are recorded. Increased values indicate worsening balance activity
Posture and spinal mobility | 6 week
  It was measured using the computer-assisted wireless Spinal Mouse device (the Spinal Mouse System, Idiag, Fehraltorf, Switzerland). The Spinal Mouse device is moved over the spine using its wheel, measuring the length of the spine, posture, and joint movements, and transferring this sequence to a computer environment. It is a reliable method that can noninvasively measure the physical characteristics and movement of the spine in a practical way. Measurements are taken from the spinous process of the seventh cervical vertebra to the third sacral vertebra. For spinal mobility, the trunk flexion posture is recorded. For postural competence values, an upright posture measurement is performed, and then a weight equal to 5% of the person's body weight is held parallel between the shoulders for 30 seconds. After the weight is still in the person's hands, the upright posture is measured again

SECONDARY OUTCOMES:
Pain level | 6 week
  Participants' pain intensity will be assessed using a visual analog scale. The scale is scored from 0 to 10, with 0 = no pain and 10 = excruciating pain.
Disability | 6 week
  OSWESTRY LOW BACK PAIN DISABILITY QUESTIONNAIRE The Oswestry Back Pain Disability Questionnaire will be used to obtain information about how much back (or leg) pain affects a person's daily activities. The questionnaire consists of 10 sections. The patient is asked to mark the most appropriate answer for themselves. The score is calculated, and the resulting percentage values are interpreted according to the values given below 0% - 20% - minimal disability 20% - 40% - moderate disability 40% - 60% - severe disability 60% - 80% - disabled 80% - 100% - bedridden

CONTACTS AND LOCATIONS:
Overall Officials: Şafak KUZU, Study Director — Kirsehir Ahi Evran Universitesi

IPD SHARING:
Plan to Share IPD: No